CLINICAL TRIAL: NCT00000906
Title: The Effect of HIV Protease Inhibitors on the Stereospecific Metabolism of Methadone in HIV-Infected Subjects
Brief Title: Interactions of HIV Protease Inhibitors and Methadone in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 401; 11357 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Methadone; HIV-1; Dose-Response Relationship, Drug; Drug Interactions; Drug Therapy, Combination; Saquinavir; Adolescent Behavior; HIV Protease Inhibitors; Ritonavir; Narcotics; Substance-Related Disorders
MeSH Terms: conditions — HIV Infections; Adolescent Behavior; Substance-Related Disorders | interventions — Ritonavir; Saquinavir; Methadone

INTERVENTIONS:
Drug: Ritonavir
Drug: Saquinavir
Drug: Methadone hydrochloride

SUMMARY:
The purpose of this study is to see if it is safe to combine methadone with two HIV protease inhibitors (PIs), ritonavir (RTV) and saquinavir (SQV), in HIV-infected patients not currently taking PIs. This study will measure the interactions between methadone and the PIs.

Methadone is used treat addicts and to treat severe pain. In order to find the safest way to use methadone with PIs, it is important to evaluate how they interact.

DETAILED DESCRIPTION:
Methadone is extensively used in the maintenance treatment of addicts and in the management of severe pain. In order to use methadone with HIV protease inhibitors correctly, it is important to evaluate and quantify interactions between the protease inhibitors and methadone.

Patients receive their usual daily dose of methadone followed with ritonavir and saquinavir, respectively, twice a day. Patients are evaluated on Day 4 for safety and tolerance, and their ritonavir dose is increased. On Day 8 patients are evaluated for a steady-state level of methadone. After 2 weeks of the protease inhibitor therapy, they return for methadone pharmacokinetic sampling at Day 15 over 24 hours. Both protease inhibitors and methadone are administered on Day 15 on an inpatient basis. On Day 30, patients are assessed for safety and tolerance.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive and have an HIV RNA count below 100,000 copies/ml within 30 days prior to study entry.
* Are taking methadone.
* Are at least 18 years old.
* Are within 40% of your ideal body weight and weigh at least 99 lbs.

Exclusion Criteria

You will not be eligible for this study if you:

* Are allergic to or are unable to take RTV or SQV.
* Have a history of treatment failure with indinavir, RTV, or SQV.
* Have a history of certain illnesses that might prevent you from completing the study.
* Have severe diarrhea or other stomach problems.
* Have taken any PI within 4 weeks prior to study entry.
* Would be unable to complete the study due to alcohol or drug abuse.
* Are co-enrolled in other protocols that have you taking medications that are prohibited in this study.
* Are taking PIs other than RTV or SQV.
* Are receiving certain therapies or are taking certain medications, including experimental drugs.
* Have an active opportunistic (AIDS-related) infection or disease that requires medication within 14 days prior to study entry.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Study Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John G. Gerber, Study Chair; Joseph Gal, Study Chair
Locations (7):
- United States (7):
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York

REFERENCES:
- [Background] Gerber JG, Rosenkranz S, Segal Y, Aberg J, D'Amico R, Mildvan D, Gulick R, Hughes V, Flexner C, Aweeka F, Hsu A, Gal J; ACTG 401 Study Team. Effect of ritonavir/saquinavir on stereoselective pharmacokinetics of methadone: results of AIDS Clinical Trials Group (ACTG) 401. J Acquir Immune Defic Syndr. 2001 Jun 1;27(2):153-60. doi: 10.1097/00126334-200106010-00010. PMID 11404537